CLINICAL TRIAL: NCT05353270
Title: Effects of Yoga on Pressor and Endothelial Function in Responses to Sodium Loading in African American Adults
Brief Title: Effects of Yoga on Sodium-induced Pressor Responses in African American Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Principal Investigator, Stacy Hunter, Assistant Professor, Texas State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7620
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Salt sensitivity
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Yoga sessions (35 minutes each) will be performed 5 times weekly for 4 weeks.
  Interventions: Behavioral: Yoga
- Waitlist control (Other): Waitlisted participants will maintain their normal diet and exercise patterns for 4 weeks prior to rerandomization to the yoga group.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Yoga — Yoga sessions will be completed 5 times per week for 4 weeks.
  Arms: Yoga
Behavioral: Waitlist control — Waitlisted participants will maintain their normal exercise and diet for 4 weeks. After follow up testing at week 4, participants will be rerandomized to the yoga condition.
  Arms: Waitlist control

SUMMARY:
This investigation aims to determine the effects of a 4-week yoga intervention on sodium-induced pressor and endothelial function responses as well as markers of renal sodium handling in African American adults.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Adults ages 18-60 years

Exclusion Criteria:

* pregnancy or within 60 days postpartum
* having taken blood pressure (including diuretics beta-blockers, ACE inhibitors, angiotensin receptor blockers, and calcium channel blockers) or statin medications within the past 3 months (statins have been demonstrated to reduce oxidative stress which could impact flow-mediated dilation);
* infection (viral or other) within the past 4 weeks;
* having adrenal or endocrine tumors (these could impact BP);
* renal disease defined as a glomerular filtration rate (GFR) of less than 60 (creatinine will be tested at initial screening and GFR will be calculated);
* prior myocardial infarction; vii) known coronary heart disease;
* personal history of stroke;
* heart failure;
* cardiac arrhythmias;
* chronic obstructive pulmonary disease;
* recent chest pain or dyspnea;
* orthopedic limitations that preclude the execution of yoga postures;
* current insulin dependence;
* currently taking steroid medications;
* currently undergoing chemotherapy or radiation;
* having practiced yoga or yogic breathing techniques at least once weekly consistently within the past 3 months;
* heat intolerance or electrolyte imbalances (hypo- or hyper-natremia or hypo- or hyper-kalemia).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from low- to high-sodium dietary conditions | Measurements will be completed after 3 days of low and 3 days of high sodium intake at baseline and after 4 weeks for both conditions.
  Blood pressure will be measured after 3 days of very low sodium and 3 days of high sodium intake.
Change in endothelial function from low- to high-sodium dietary conditions. | Measurements will be completed after 3 days of low- and 3 days of high-sodium intake at baseline and at week 4.
  Flow-mediated dilation will be measured via ultrasound imaging of the upper arm after 3 days of low- and 3 days of high- sodium dietary conditions.
Change in arterial stiffness from low- to high-sodium dietary conditions. | Measurements will be completed after 3 days of low- and 3 days of high-sodium intake at baseline and at week 4.
  Cardio-ankle vascular index will be measured after 3 days of low- and 3 days of high-sodium intake.

SECONDARY OUTCOMES:
Change in urinary sodium excretion from low- to high-sodium dietary conditions. | Measurements will be completed after 3 days of low- and 3 days of high-sodium intake at baseline and at week 4.
  24-hour urine collection will be completed after 3 days of low- and after 3 days of high-sodium dietary conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Physiology Laboratory-Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hunter SD, Kavouras SA, Rahimi M. Exploring heated exercise as a means of preventing the deleterious effects of high-sodium intake in Black women. Am J Physiol Heart Circ Physiol. 2023 Jun 1;324(6):H833-H839. doi: 10.1152/ajpheart.00699.2022. Epub 2023 Apr 7. PMID 37027326